CLINICAL TRIAL: NCT05227274
Title: Reliability Study of a Motor Function Measure Digitalized Playful Completion Modules
Acronym: MFM-Play
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1088
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Neuromuscular Diseases
Keywords: Motor Function Assessment; Reliability study; Patient Participation
MeSH Terms: conditions — Neuromuscular Diseases; Patient Participation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MFM-Play: Neuromuscular disease patients completed MFM using MFM-Play
  Interventions: Other: Items completion with or without a MFM-Play

INTERVENTIONS:
Other: Items completion with or without a MFM-Play — Patients will completed 3 MFM during the follow-up, two times using the MFM-Play, and one without the MFM-Play Delay between each MFM completion will be 1 month ± 15 days

SUMMARY:
Neuromuscular diseases include more than 200 rare disorders affecting muscles or the nervous system. Functional scales assessing motor function are tools allowing to measure the evolution of motor impairment of patients with a neuromuscular disease. They are frequently used as main outcome measures in clinical trials which are currently in full development thanks to advances in genetic and drug researches.

Among the available scales, the Motor Function Measure (MFM), a scale consisting of 32 items, had shown good metrological properties in terms of validity, reliability and sensitivity to change, regardless of the diagnosis and extent of motor impairment.

By exploring the potential of digital technologies applied to MFM, investigators created a completion module composed of animations with different playful and informative scenarios displayed on a digital tablet.

The main purpose of this project is to conduct a multicentre study to assess reliabilities of the MFM completed using the MFM-Play.

Expected benefits of this project are to improve the experience and the participation of the children to who is often imposed multiple assessments during the numerous follow-up visits of clinical trials, while maintaining good metrological properties of the MFM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a neuromuscular disease confirmed by the clinic, electroneuromyography (ENMG), biology, muscular biopsy, or genetic
* aged ≥ 2 yo and ≤ 60 yo
* having been informed and not objecting to participating in the study (information and non-opposition of parents/holders of parental authority for minor patients)

Exclusion Criteria:

* participating in other interventional research with an exclusion period that is still ongoing or that may interfere with the results of this study
* having had surgery or illness impacting their motor function within the last 6 months
* having understanding and/or behavioral deficiencies preventing rigorous assessment
* Patient placed under legal protection (this includes guardianship, curatorship and safeguard of justice)

Ages: 2 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with a follow-up in a French neuromuscular reference center
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Comparison of item scoring between 2 MFM completion. | 3 months
  Level of agreement between MFM item scores reported by physiotherapists during 2 different MFM completion using the MFM-Play.
  Level of agreement between MFM item scores reported by a same physiotherapist during a MFM completion using the MFM-Play and a MFM completed conventionally.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Centre de référence maladies neuromusculaires Hôpital Morvan - CHRU de Brest, Brest
  - Service de Rééducation Fonctionnelle Pédiatrique - L'Escale - Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron
  - Service de Médecine Physique et de Réadaptation Pédiatrique Hôpital Couple-Enfant CHU de Grenoble, La Tronche
  - Centre de référence maladies neuromusculaires Hôpital Salengro CHU Lille, Lille
  - Consultation pluridisciplinaire MNM adulte Hôpital de la Croix Rousse, Groupement Hospitalier Nord HCL, Lyon
  - ESEAN - APF France Handicap, Nantes
  - Consultation de pédiatrie- maladie neuromusculaire Hôpital Armand Trousseau APHP, Paris
  - Service de Médecine Physique et de Réadaptation Pédiatrique Hôpital Bellevue CHU Saint Etienne, Saint-Etienne
  - Centre de référence MNM Adulte Saint Etienne - service neurologie CHU Hôpital Nord, Saint-Priest-en-Jarez
  - Centre de référence des maladies neuromusculaires enfants Hôpital des enfants CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No